CLINICAL TRIAL: NCT05447117
Title: Subthreshold Micropulse 532 nm Green Laser Treatment of Acute Central Serous Chorioretinopathy: 18-month Results
Brief Title: Subthreshold Micropulse Laser Treatment of Acute Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosny Ahmed Zein, Assistant Professor, Minia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCR2019
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acute Central Serous Retinopathy With Subretinal Fluid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Micropulse laser — 532 nm green subthreshold micropulse laser (GSML) as a treatment for acute central serous chorioretinopathy (CSCR).

SUMMARY:
To evaluate the efficacy and safety of 532 nm green subthreshold micropulse laser (GSML) as a treatment for acute central serous chorioretinopathy (CSCR).

DETAILED DESCRIPTION:
This prospective study included 42 eyes of 42 patients with acute CSCR treated with IRIDEX™ IQ 532 nm GSML. The study was conducted at Minia University Hospital and Genaidy Ophthalmology Center, Minia, Egypt between October 2019 and May 2022. All patients were subjected to a complete ophthalmological examination, fluorescein angiography (FA) and optical coherence tomography (OCT) at baseline and each follow-up visit 1, 3 and 18 months after laser treatment

ELIGIBILITY:
Inclusion Criteria:

* acute CSCR

Exclusion Criteria:

* chronic CSCR Previously treated case of Acute CSCR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change in visual acuity | 18 months
  resolution of subretinal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No